CLINICAL TRIAL: NCT07116928
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study of the Effects of Ganagliflozin on the Progression of Kidney Disease in Subjects With Type 2 Diabetes Mellitus and Chronic Kidney Disease
Brief Title: Ganagliflozin on the Progression of Kidney Disease in Subjects With Type 2 Diabetes Mellitus and Chronic Kidney Disease
Acronym: GLOW-CKD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HDHYJ-LC-2
Record Dates: First submitted 2025-07-23; First posted 2025-08-12 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-08

CONDITIONS: T2DM (Type 2 Diabetes Mellitus); CKD - Chronic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ganagliflozin (Experimental): 50 mg Once daily, 120 weeks
  Interventions: Drug: ganagliflozin
- placebo (Placebo Comparator): 50 mg Once daily, 120 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ganagliflozin — 50 mg Once daily, 120 weeks
  Arms: ganagliflozin
Drug: Placebo — 50 mg Once daily, 120 weeks
  Arms: placebo

SUMMARY:
This study aims to investigate the impact of adding Ganagliflozin tablets to the current background therapy on preventing the progression of kidney disease in subjects with type 2 diabetes and chronic kidney disease. The efficacy and safety will be evaluated by comparing the effects of Ganagliflozin tablets and placebo tablets added to the current background treatment over 120 weeks

DETAILED DESCRIPTION:
A phase IV clinical study on the efficacy and safety of Ganagliflozin in treating patients with type 2 diabetes and chronic kidney disease (multicenter, randomized, double-blind, placebo parallel controlled). 1244 subjects all received a stable dose of ACEi or ARB for at least 4 weeks before enrollment.

Efficacy assessment: Compared with the placebo group, time to the first occurrence of kidney disease progression and the changes in eGFR slope, UACR, and score of KDQOL-36 were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals aged 18 years and above;
* Meets the diagnostic criteria for T2DM;
* Meets the diagnostic criteria for CKD, during the screening period（CKD-EPI Formula）: eGFR ≥ 30 to < 60 mL/min/1.73m^2, and UACR is ≥ 30 to < 5000 mg/g; Or eGFR ≥ 60 to < 90 mL/min/1.73m^2, and UACR is ≥ 300 to < 5000 mg/g ;
* HbA1c ≥ 6.5% to ≤ 12%;
* If there are no contraindications or special instructions, all subjects must take a stable dose of ACEi or ARB at least 4 weeks before randomization;

Exclusion Criteria:

* Patients with type 1 diabetes or other special types of diabetes;
* A medical history or clinical evidence indicating that the subjects have other primary kidney diseases and secondary kidney diseases other than type 2 diabetes (including but not limited to lupus nephritis, ANCA-related nephritis);
* History of kidney transplantation;
* Blood potassium level > 5.5 mmol/L during the screening period.
* New York Heart Association (NYHA) classification of grade IV during the screening period;
* Experienced ketoacidosis, myocardial infarction, unstable angina pectoris, stroke, transient ischemic attack (TIA), hospitalization due to heart failure, or hospitalization due to urinary tract infection or acute kidney injury within 12 weeks before the screening period;
* Receiving ACEi and ARB in combination;
* Receiving mineralocorticoid receptor antagonists (MRA) or direct renin inhibitors (DRI) within 8 weeks before randomization;
* Receiving drugs with immunosuppressive effects (such as cyclophosphamide, cyclosporine A, tacrolimus, etc.) or biological agents (rituximab, belimumab, etc.) during the 12 weeks before the screening period;
* Receiving SGLT-2 inhibitors or GLP-1 receptor agonists within 8 weeks before the screening, or have previously used SGLT-2 inhibitor drugs and discontinued due to poor efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1244 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2031-10-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
The average change in eGFR as measured by the total slope of eGFR from baseline to week 120 | Baseline to Week 120

SECONDARY OUTCOMES:
Time to the first occurrence of kidney disease progression | from baseline to Week 120
  The progression of kidney disease is defined as:
  1. maintenance dialysis or
  2. receipt of a kidney transplant or
  3. sustained decline in eGFR to < 15 mL/min/1.73m^2 or
  4. a sustained decline of ≥ 40% in eGFR from baseline or
  5. doubling of serum creatinine or
  6. renal death
The proportion of subjects with a total slope of eGFR greater than -3 mL/min/1.73 m²/year from baseline to week 120 | from baseline to week 120
The average change in eGFR as measured by the total slope of eGFR from baseline to week 2 and week 8，from week 2 and week 8 to week 120 | from baseline to week 2 and week 8，from week 2 and week 8 to week 120
The changes in urine albumin-to-creatinine ratio (UACR) at each visit compared to the baseline | from baseline to week 120
Changes in the scores of the Kidney Disease Quality of Life-36 Scale (KDQOL-36) compared to the baseline | from baseline to week 120
  The higher the score, the better the patient's quality of life related to CKD
Changes in the scores of the European Five-Dimensional Health Scale (EQ-5D-5L) compared to the baseline | from baseline to week 120
  Higher the score means the better quality of life

OTHER OUTCOMES:
time to the first occurrence of cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, or hospitalization for heart failure | from baseline to week 120
Changes in liver stiffness measurement (LSM) of liver transient elastography | from baseline to week 52 and 120
change in the staging of diabetic retinopathy measured by non-mydriatic fundus photography | from baseline to week 52 and 120
Changes in control attenuation index (Cap) of liver transient elastography | from baseline to week 52 and 120

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai sixth People's Hospital, Shanghai, Shanghai Municipality, China